CLINICAL TRIAL: NCT01716000
Title: Optical Imaging and User Perception Study of Vaginal Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); ImQuest Pharmaceuticals, Inc. (Industry); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00038440; U19AI077289 (NIH)
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Characterize Gel Distribution in the Vagina; Study Women's Sensory Perceptions and Preferences of Gel
Keywords: vaginal gel; vaginal coating; sensory perceptions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 mL vaginal gel (Experimental): 2 mL gel inserted vaginally for completion of vaginal gel imaging and computer aided self interview.
  Interventions: Other: vaginal gel imaging; Behavioral: computer aided self interview
- 4 mL vaginal gel (Experimental): 4 mL gel inserted vaginally for completion of vaginal gel imaging and computer aided self interview.
  Interventions: Other: vaginal gel imaging; Behavioral: computer aided self interview

INTERVENTIONS:
Other: vaginal gel imaging — Imaging of vaginal gel distribution using two investigational techniques (low coherence interferometry and fluorimetry).
Behavioral: computer aided self interview — Questionnaire to gather the perceptions and preferences of the subject with respect to the vaginal gel.

SUMMARY:
This study will compare two investigational techniques for measuring how vaginal gels spread and coat the vagina. This study will also explore the experiences and opinions of women using this vaginal gel. We want to understand how the characteristics of a gel, such as a gel's thickness or consistency, affect how the gel spreads and feels in the body. We hope to use the information we learn from this study to develop future vaginal gels that could be combined with medications and used to slow down or stop the spread of sexually transmitted infections.

DETAILED DESCRIPTION:
The pharmacokinetics of a microbicide gel, i.e. the time- and space-dependent distribution of its active microbicidal ingredient(s) (APIs) throughout the body, derives from the time- and space-dependent distribution of the gel itself within the vaginal canal. That distribution may also serve as a physical barrier that retards migration of semen-borne HIV virions to epithelial surfaces. Within the vagina, the gel creates local physical forces ("stresses") against the epithelial surfaces; and its distribution along the canal might be so extensive that gel leaks out from the introitus. A woman may have sensations of those stresses and also feel gel leakage. Thus, intravaginal microbicide gel distribution is central to both its biological functioning (to deliver APIs and also to slow HIV transport) and the behavioral perception of it by users (i.e. how it "feels" and whether that experience is pleasurable or not). The latter, in turn, can govern acceptability of the gel and adherence to designated gel use in clinical trials. This study will characterize and correlate gel distribution and women's sensory perceptions and preferences of that distribution, for two relevant volumes (2 mL and 4 mL) of a current microbicide placebo gel. An optical vaginal imaging device will measure gel distribution in the vagina. A computer-assisted self-interview (CASI) survey will capture women's perceptions and preferences.

ELIGIBILITY:
Inclusion Criteria:

* have had vaginal penetrative intercourse within the last 12 months
* have a regular menstrual cycle (between 24-35 days) and be able to record the day of onset of menses in a menstrual diary
* able to ambulate for 20 consecutive minutes after vaginal self-insertion of gel using an applicator
* willing to use a condom when engaging in sexual intercourse within 4 days before a study visit
* willing to avoid using any mechanical sex toy within 1 day before a study visit
* willing to use one of the following contraception methods if engaging in sexual intercourse during the length of participation in the study (hormonal contraceptive, tubal ligation, non-surgical procedure such as permanent transcervical sterilization, Fallopian tubes removed, partner vasectomy)
* able to provide informed consent

Exclusion Criteria:

* pregnant, potentially pregnant, nursing, or trying to conceive
* allergic to latex, fluorescein, hydroxyethylcellulose, ascorbic acid, sodium citrate, citric acid
* using an intrauterine device (IUD)
* using depo-provera
* douching during the course of participation in the study
* had medical or cosmetic surgery involving the reproductive organs or genitals within the past 6 months
* have a gynecological infection or other condition requiring treatment, such as candidiasis, chlamydia trachomatis, trichomoniasis, HIV, herpes simplex virus (HSV), neisseria gonorrhea, symptomatic bacterial vaginosis, or syphilis
* currently enrolled in any other research studies involving the application of vaginal formulations
* employed or supervised by the study investigators
* have any other condition that, in the opinion of the study physician, would contraindicate participation in the study

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
number and frequency of adverse events | up to 6 months

SECONDARY OUTCOMES:
extent of vaginal gel coating | at imaging visit 1 (between 1-6 weeks after enrollment) and at imaging visit 2 (between 1 - 6 weeks after imaging visit 1)
  extent of vaginal gel coating is measured by: algebraic and harmonic mean gel thickness, total vaginal surface area with detectable gel coating, fraction of total vaginal surface area containing detectable gel coating, linear extent of gel coating along the vaginal canal, ratio of linear extent of coating to the length of the vaginal canal
uniformity of vaginal gel coating | at imaging visit 1 (between 1-6 weeks after enrollment) and at imaging visit 2 (between 1 - 6 weeks after imaging visit 1)
  uniformity of vaginal gel coating is measured by: coefficient of variation of local coating thickness and the number, location, and sizes of individual bare spots of uncoated vaginal surface within the overall gel coating envelope
subject perception and preference of vaginal gel | at imaging visit 1 (between 1-6 weeks after enrollment) and at imaging visit 2 (between 1 - 6 weeks after imaging visit 1)
  responses to the computer aided self interview questions, grouped into the following scales: Leaks with Application, Ease of Application, Portability, Intravaginal Feel, Perception of Leakage with Ambulation, Leaking with Ambulation, Leakage Across Time, Sticky with Ambulation, Perception of Natural Wetness, and Lubrication Moisture on Ambulation.

CONTACTS AND LOCATIONS:
Overall Officials: David F. Katz, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States